CLINICAL TRIAL: NCT02548988
Title: Immediate Effect of Selective Neuromuscular Electrical Stimulation of Vastus Medialis Obliquus in Women With Patellofemoral Pain Syndrome
Brief Title: Selective Neuromuscular Electrical Stimulation on VMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 056711/2015
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Patellofemoral Pain Syndrome; Electric Stimulation
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy (Experimental): Healthy women are submitted to selective neuromuscular electrical stimulation on VMO.
  Interventions: Other: Neuromuscular Electrical Stimulation
- Patellofemoral pain syndrome (Experimental): Women with patellofemoral pain syndrome are submitted to selective neuromuscular electrical stimulation on VMO.
  Interventions: Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — Selective Neuromuscular Electrical Stimulation on VMO

SUMMARY:
The purpose of this study is analyze the immediate effect of selective neuromuscular electrical stimulation of vastus medialis obliquus (VMO) in the electrical activity of VMO and vastus lateralis (VL) and in the isokinetic performance of women with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy group:
* with no history of osteomyoarticular lesion or surgery in the lower limbs in the previous six months
* non-corrected neurological, vestibular, visual and/or hearing impairment
* For Patellofemoral pain syndrome group:
* clinical diagnosis of patellofemoral pain syndrome
* absence of other disorders in the knee
* refer pain at leafs two of the following activities: when remain seated for a long period, squat, kneel and go up or down stairs.

Exclusion Criteria:

* Individuals experiencing pain during collection procedures
* do not perform exercises as instructed by the researches

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity (root mean square - RMS) of vastus medialis obliquus | Change from baseline in Electromyographic activity at 30 minutes
  The immediate effect of neuromuscular electrical stimulation will be measured through surface electromyography and the variable analyzed will be root mean square (RMS).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil